CLINICAL TRIAL: NCT03956030
Title: Effect of Formal Contraception Handouts on Postpartum Birth Control Use and Methods
Brief Title: Effect of Formal Contraception Handouts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient research staff to recruit and complete study.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christina DeAngelis, Assistant Professor Women's Health Division, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00012248
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Contraception; Counseling
Keywords: Female Contraception; Education

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in which the intervention group will receive an educational handout on contraception and the control group will receive a handout on nutrition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive educational handout on contraception.
  Interventions: Other: Contraception Handout
- Control (Experimental): Control group will receive educational handout on nutrition.
  Interventions: Other: Nutritional Handout

INTERVENTIONS:
Other: Contraception Handout — Handout covering contraception options
  Arms: Intervention
Other: Nutritional Handout — Handout covering nutrition
  Arms: Control

SUMMARY:
The hypothesis of this study is to determine if distribution of a standardized educational handout on contraceptive options given to patients in the prenatal office setting will increase contraception use six months postpartum.

DETAILED DESCRIPTION:
Reducing unintended pregnancies and those that are conceived within 18 months of a previous livebirth is an important health concern in the United States. Both unintended and close-interval pregnancies constitute 40% and 35% of pregnancies in the United States respectively with some overlap between the two categories and are associated with adverse maternal and fetal outcomes. A national survey found that 17.8% of women using 'less-effective' methods and 23% of women using no birth control became pregnant in ≤18 months2. Access to better contraception education could potentially decrease the proportion of unintended pregnancies and close-interval pregnancies. In addition to the health concerns, 58% of women in the US would like more information about contraceptive options, and organized handouts on birth control have been shown to contribute to the choice in birth control. However, there has been conflicting evidence about which educational methods increase postpartum contraception use. Therefore, the investigators propose a randomized controlled trial (RCT) that assesses whether a handout on contraception options increases postpartum birth control use. The control group would receive a nutrition handout, and the intervention group would receive a handout on birth control options in addition to each receiving the standard of care. The researchers would also give pre- and post-natal questionnaires, covering patient satisfaction, intention to use birth control, and how often a provider discusses birth control options.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are pregnant and are 24-28 weeks gestational age at the time of recruitment
2. Women >18 years of age
3. Women with low-risk pregnancies

Exclusion Criteria:

1. Women who receive prenatal care by the Maternal Fetal Medicine department for high-risk pregnancies
2. Women who are members of an at-risk population including any women who is a prisoner, cannot provide consent, or is <18 years of age
3. Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will recruit women who are 24-28 weeks gestational age.
Enrollment: 8 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina DeAngelis, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Women's Health Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 4 | 4
Completed | 1 | 1
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (6.9) | 27.0 (5.1) | 27.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Contraception Use
Description: Participants were sent a survey electronically at 8 weeks which asked the question "Now that you have delivered, are you currently using birth control? (yes or no)" The data table reflects the number who answered YES and the number who answered NO to this question per group.
Time Frame: 8 weeks postpartum
Population: Subjects who completed the 8 week survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 2
Participants
  Reported YES to contraception use | 1 | 1
  Reported NO to contraception use | 0 | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Termination of the study leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03956030/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT03956030/ICF_001.pdf